CLINICAL TRIAL: NCT01815294
Title: A Pivotal Bioequivalence Study of DOXIL/CAELYX Manufactured at a New Site in Subjects With Advanced or Refractory Solid Malignancies Including Subjects With Ovarian Cancer.
Brief Title: A Pivotal Bioequivalence Study of DOXIL/CAELYX (Doxorubicin HCL) in Patients With Advanced or Refractory Solid Malignancies Including Patients With Ovarian Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR100961; DOXILNAP1002 (Other: Janssen Research & Development, LLC); 2013-000376-15 (EudraCT Number)
Record Dates: First submitted 2013-03-14; First posted 2013-03-21 (Estimated); Last update posted 2015-12-04 (Estimated); Status verified 2015-12

CONDITIONS: Neoplasms; Neoplasms, Ovarian; Neoplasms, Breast; Advanced or Refractory Solid Malignancies
Keywords: Ovarian cancer; Breast cancer; Solid malignancy; Advanced or refractory solid malignancy; Metastatic cancer; DOXIL/CAELYX; Doxorubicin HCL; Bioequivalence
MeSH Terms: conditions — Neoplasms; Ovarian Neoplasms; Breast Neoplasms; Neoplasm Metastasis | interventions — liposomal doxorubicin; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment A: DOXIL/CAELYX (doxorubicin) (Experimental): 50 mg/m2 of doxorubicin manufactured at the current site of manufacturing administered by IV infusion over 90 minutes on Day 1
  Interventions: Drug: DOXIL/CAELYX (doxorubicin) Treatment Sequence AB; Drug: DOXIL/CAELYX (doxorubicin) Treatment Sequence BA
- Treatment B: DOXIL/CAELYX (doxorubicin) (Experimental): 50 mg/m2 of doxorubicin manufactured at the new site of manufacturing (test product) administered by IV infusion over 90 minutes on Day 1
  Interventions: Drug: DOXIL/CAELYX (doxorubicin) Treatment Sequence AB; Drug: DOXIL/CAELYX (doxorubicin) Treatment Sequence BA

INTERVENTIONS:
Drug: DOXIL/CAELYX (doxorubicin) Treatment Sequence AB — Cycle 1 = Treatment A, Cycle 2 = Treatment B
Drug: DOXIL/CAELYX (doxorubicin) Treatment Sequence BA — Cycle 1 = Treatment B, Cycle 2 = Treatment A

SUMMARY:
The purpose of this study is to support the qualification of a replacement manufacturing site for DOXIL/CAELYX (doxorubicin HCL).

DETAILED DESCRIPTION:
This is a randomized (individuals will be assigned in a random order to study treatment sequences), open-label (identity of assigned treatment sequences will be known), single dose, 2-cycle, crossover (patients will receive both treatments in a random order) bioequivalence study of DOXIL/CAELYX (doxorubicin HCL) in patients with advanced or refractory solid malignancies (including patients with ovarian cancer). This study has an adaptive 2-stage design. Bioequivalence based on encapsulated doxorubicin will be tested at the end of Stage 1 using data from at least 24 ovarian cancer patients. An interim analysis of free doxorubicin will be performed at the end of Stage 1 using data from 42 patients of all cancer types. The study may continue into Stage 2 with additional patients of all cancer types; and final evaluation of bioequivalence for free doxorubicin will be performed at the end of Stage 2. The study will include a screening phase followed by an open-label treatment phase consisting of 2 doxorubicin treatment cycles and an end-of-treatment visit on Cycle 3, Day 1. Participants may enter an optional extension phase after 2 cycles. Safety will be monitored throughout the study. Blood samples for pharmacokinetic analysis will be obtained from all participants at specified times over 29 days after starting each study drug administration in Cycles 1 and 2 for determination of plasma concentrations of encapsulated and free doxorubicin.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with advanced or refractory solid malignancies: histologically or cytologically confirmed advanced ovarian cancer failing platinum-based chemotherapy; histologically or cytologically confirmed metastatic breast cancer after failing approved life-prolonging therapies; any histologically or cytologically confirmed solid malignancy that is metastatic or unresectable, and for which standard treatment is no longer an option
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Recovered from acute toxicity of any prior treatment (exemptions: alopecia, grade-1 neuropathy)
* Prior doxorubicin (or other anthracyclines) at cumulative dose of <=360 mg/m2 or cumulative epirubicin dose <=720 mg/m2 (calculated using doxorubicin equivalent doses: 1 mg doxorubicin = 1 mg DOXIL/CAELYX = 0.3 mg mitoxantrone = 0.25 mg idarubicin)
* Adequate liver, bone marrow, and renal function according to protocol-defined parameters
* Left ventricular ejection fraction (LVEF) within normal limits of the institution as determined by multiple uptake gated acquisition (MUGA) or echocardiography
* Agrees to protocol-defined use of effective contraception
* Negative pregnancy test at screening (applicable to women of child bearing potential) within 7 days prior to starting treatment

Exclusion Criteria:

* Positive history of known brain metastases or leptomeningeal disease (patients with brain metastases can only be enrolled if the following conditions are all met: treated and stable for >4 weeks [>2 weeks after SRS/Cyberknife]; no evidence for progression or hemorrhage after treatment; steroid treatment discontinued at least 2 weeks prior to first administration of doxorubicin; enzyme inducing anti-epileptic drugs discontinued at least 4 weeks before first administration of doxorubicin
* History of hypersensitivity reaction to doxorubicin HCl or other components of DOXIL/CAELYX
* Any major surgery, radiotherapy, or immunotherapy within the last 21 days (limited palliative radiation allowed >=2 weeks prior to the first dose; >=4 weeks for whole brain radiotherapy); chemotherapy regimens with delayed toxicity within the last 4 weeks (or within the last 6 weeks for prior nitrosourea or mitomycin C); chemotherapy regimens given continuously or on a weekly basis with limited potential for delayed toxicity within the last 2 weeks
* Use of an investigational drug within 21 days or 5 half-lives (whichever is shorter) prior to the first dose of doxorubicin
* Unstable angina or myocardial infarction within the preceding 12 months; congestive heart failure or any history of uncontrolled cardiac disease >Class II based on New York Heart Association Criteria
* Has an infection that is either an uncontrolled infection, clinically important (occurred within 4 weeks prior to first dose of study agent), or requiring current systemic intravenous treatment
* Uncontrolled concurrent illness including, but not limited to, poorly controlled hypertension or diabetes, or psychiatric illness/social situation that may potentially impair patient's compliance with study procedures
* Concomitant use of strong CYP3A4 inhibitors (such as clarithromycin, diltiazem, erythromycin, itraconazole, ketoconazole, nefazodone, ritonavir, telithromycin and verapamil) and strong CYP3A4 inducers (such as carbamazepine, phenobarbital, phenytoin, rifampin and St John's wort) from at least 4 weeks before the first dose of doxorubicin in Cycle 1 and until after completion of all pharmacokinetic sampling in Cycle 2
* Has any condition that, in the opinion of the investigator, would make participation not be in the best interest (eg, compromise the well-being) of the patient or that could prevent, limit, or confound the protocol-specified assessments
* Woman who is pregnant, or breast-feeding, or planning to become pregnant or is a man who plans to father a child while enrolled in this study or within 3 months after the last dose of study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2013-05; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration of encapsulated doxorubicin in participants with ovarian cancer | Predose Day 1 Cycles 1-2; Postdose Cycles 1-2 at 15 min, 30 min, 60 min, 90 min, 95 min, 105 min, 2 h, 3 h, 4 h, 6 h, 8 h, 24 h, 48 h, 72 h, 96 h, 168 h, 336 h, 504 h, 672 h
Area under the plasma-concentration-versus time curve from time 0 to time t of encapsulated doxorubicin in participants with ovarian cancer | Predose Day 1 Cycles 1-2; Postdose Cycles 1-2 at 15 min, 30 min, 60 min, 90 min, 95 min, 105 min, 2 h, 3 h, 4 h, 6 h, 8 h, 24 h, 48 h, 72 h, 96 h, 168 h, 336 h, 504 h, 672 h
Area under the plasma-concentration-versus time curve from time 0 to infinite time of encapsulated doxorubicin in participants with ovarian cancer | Predose Day 1 Cycles 1-2; Postdose Cycles 1-2 at 15 min, 30 min, 60 min, 90 min, 95 min, 105 min, 2 h, 3 h, 4 h, 6 h, 8 h, 24 h, 48 h, 72 h, 96 h, 168 h, 336 h, 504 h, 672 h

SECONDARY OUTCOMES:
Maximum observed plasma concentration of free doxorubicin in participants with solid malignancies | Predose Day 1 Cycles 1-2; Postdose Cycles 1-2 at 15 min, 30 min, 60 min, 90 min, 95 min, 105 min, 2 h, 3 h, 4 h, 6 h, 8 h, 24 h, 48 h, 72 h, 96 h, 168 h, 336 h, 504 h, 672 h
Area under the plasma-concentration-versus time curve from time 0 to time t of free doxorubicin in participants with solid malignancies | Predose Day 1 Cycles 1-2; Postdose Cycles 1-2 at 15 min, 30 min, 60 min, 90 min, 95 min, 105 min, 2 h, 3 h, 4 h, 6 h, 8 h, 24 h, 48 h, 72 h, 96 h, 168 h, 336 h, 504 h, 672 h
Area under the plasma-concentration-versus time curve from time 0 to infinite time of free doxorubicin in participants with solid malignancies | Predose Day 1 Cycles 1-2; Postdose Cycles 1-2 at 15 min, 30 min, 60 min, 90 min, 95 min, 105 min, 2 h, 3 h, 4 h, 6 h, 8 h, 24 h, 48 h, 72 h, 96 h, 168 h, 336 h, 504 h, 672 h
Number of participants affected by adverse events by MedDRA system organ class (SOC) and Preferred term (PT) | Up to 30 days after the last dose of study medication
Response | Up to Cycle 3 Day 1
  Investigator determined response is defined by complete response, partial response or stable disease criteria

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (8):
- United States (2):
  - Nashville, Tennessee
  - San Antonio, Texas
- Belgium (2):
  - Brussels
  - Wilrijk
- Spain (3):
  - Barcelona
  - Madrid
  - Valencia
- London, United Kingdom

REFERENCES:
- See also: A Pivotal Bioequivalence Study of DOXIL®/CAELYX® Manufactured at a New Site in Subjects With Advanced or Refractory Solid Malignancies Including Subjects With Ovarian Cancer — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_7051&studyid=3629&filename=CR100961_CSR.pdf